CLINICAL TRIAL: NCT03301181
Title: A Phase 1, Open-label, Parallel-group, Fixed-sequence Study to Investigate the Effect of the CYP3A Inducer Rifampin and the CYP3A Inhibitor Itraconazole on the Pharmacokinetics of BGB-3111 in Healthy Subjects
Brief Title: Phase 1 Study to Investigate Effect of Rifampin and Itraconazole on the Pharmacokinetics of BGB-3111 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: BGB-3111-104
Record Dates: First submitted 2017-09-29; First posted 2017-10-04 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2018-06

CONDITIONS: Healthy Volunteers: Asian, Non-Asian
MeSH Terms: interventions — zanubrutinib; Rifampin; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Approximately 20 subjects to receive BGB-3111 and rifampin
  Interventions: Drug: BGB-3111 (Arm A); Drug: Rifampin
- Arm B (Experimental): Approximately 20 subjects to receive BGB-3111 and itraconazole
  Interventions: Drug: BGB-3111 (Arm B); Drug: Itraconazole

INTERVENTIONS:
Drug: BGB-3111 (Arm A) — 320 mg BGB-3111 single oral dose
  Arms: Arm A
Drug: Rifampin — 600 mg rifampin once daily
  Other Names: Rifadin, Rimactane
  Arms: Arm A
Drug: BGB-3111 (Arm B) — Up to 80 mg BGB-3111 single oral dose
  Arms: Arm B
Drug: Itraconazole — 200 mg itraconazole once daily
  Other Names: Sporanox, Orungal
  Arms: Arm B

SUMMARY:
Phase 1 study in healthy subjects to determine the effect of rifampin (Part A) or itraconazole (Part B) on the pharmacokinetics of BGB-3111

DETAILED DESCRIPTION:
This is a Phase 1 open-label, parallel-group study in healthy subjects. Subjects in Part A will receive a single dose of BGB-3111 before and during consecutive daily doses of strong cytochrome P450 CYP3A inducer, rifampin, to investigate its effect on the pharmacokinetics of BGB-3111. Following an interim data analysis, subjects in Part B will receive a single dose of BGB-3111 before and during consecutive daily doses of strong CYP3A inhibitor, itraconazole, to investigate its effect on the pharmacokinetics of BGB-3111.

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index (BMI)18 - 32 kg/m2, inclusive.
2. Subjects of Asian (first- or second-generation) and non-Asian descent.
3. In good general health as assessed by the Investigator.
4. Females must be nonpregnant and nonlactating, and females of childbearing potential will agree to use required contraception.
5. Males without a vasectomy will agree to use required barrier contraception, and will agree to not donate sperm from the time of the first dose of BGB-3111 until ≥90 days after the last dose of BGB-3111.Able to comprehend and willing to sign consent.

Exclusion Criteria:

1. Subjects with a clinically relevant history or presence of any clinically significant disease.
2. Evidence of bacterial, viral, fungal, parasitic infections within 4 weeks prior to the first dose of study drug.
3. History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance.
4. History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs.
5. History of alcoholism or drug/chemical abuse within prior year.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2017-11-07 (Actual); Study Completion 2017-11-13 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of BGB-3111 and rifampin to evaluate protocol specified PK parameters | Part A: Days 1 and 10
Plasma concentration of BGB-3111 and itraconazole to evaluate protocol specified PK parameters | Part B: Days 1 and 6

SECONDARY OUTCOMES:
Safety as assessed by adverse events | Part A: up to 19 days: Part B: up to 14 days
Safety as assessed by electrocardiogram (ECG) measurements | Part A: Days 1 and 10, from screening to end of study visit; up to Day 19; Part B: Days 1 and 6, from screening to end of study visit; up to Day 14

CONTACTS AND LOCATIONS:
Overall Officials: William Novotny, MD, Study Director — BeiGene
Locations (1):
- West Coast Clinical Trials (WCCT), Cypress, California, United States